CLINICAL TRIAL: NCT05163158
Title: CENtral Blood Pressure Targeting: a Pragmatic RAndomized Pilot TriaL in Advanced Chronic Kidney Disease
Acronym: CENTRAL-CKD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Remi Goupil, MD MSc, Principal Investigator, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CENTRAL-CKD Protocol Version 1
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chronic Kidney Diseases; Hypertension
Keywords: Central blood pressure; Central hypertension; Chronic kidney disease; Hypertension; Arterial stiffness
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Central BP target (Experimental): Participants randomized to central BP target will be treated with anti-hypertensive agents to achieve a clinic central SBP < 130 mmHg.
  Interventions: Other: Central vs brachial systolic blood pressure targeting
- Brachial BP target (standard of care) (Active Comparator): Participants randomized to a brachial BP target will be treated with anti-hypertensive drugs to achieve a clinic brachial SBP <130 mmHg.
  Interventions: Other: Central vs brachial systolic blood pressure targeting

INTERVENTIONS:
Other: Central vs brachial systolic blood pressure targeting — Participants will be randomized to either a central BP target (intervention) or a brachial BP target (standard care). For each group, the source of the BP (central or brachial) will be blinded and only the BP values will be provided to the attending Nephrologist. In both cases, the target SBP will be <130 mmHg.

SUMMARY:
Background: Emerging data favors aortic blood pressure (BP) over brachial cuff BP in predicting CV and renal complications, as this BP directly impacts the heart, brain and kidneys. In parallel, central BP measuring devices have been developed that are more accurate towards aortic BP and easy to use without training. In no other condition than advanced chronic kidney disease (CKD) is BP control as important, since undertreatment is associated with adverse CV events and progression towards end-stage kidney disease (ESKD), while overtreatment similarly leads to adverse CV events and injurious falls but also acute kidney injury which can precipitate ESKD. To this day, standard BP management relies on brachial cuff BP, which is an imprecise surrogate marker of aortic BP, more so in the advanced CKD population. Considering that these patients have a high risk of CV morbidity and mortality and is a group where brachial BP may be the least reliable, it can be beneficial to manage hypertension in this population using central BP measurements. With the development of affordable and easy to use central BP devices, routine use of central BP in hypertension would now become a reality. However, the superiority of central BP to traditional brachial cuff BP in regard to clinical outcomes will first need to be demonstrated.

Objectives: To demonstrate that targeting central BP in advanced CKD patients as opposed to brachial cuff BP is feasible and results in lower arterial stiffness after 12 months of follow-up.

Methods: The CENTRAL-CKD trial is an investigator-initiated prospective parallel-group 1:1 randomized double-blinded multicenter pragmatic pilot trial. Patients with CKD stages 4 and 5 (n=116) will be randomized to either a central systolic BP target < 130 mmHg (intervention) or brachial systolic BP target < 130 mmHg (standard care). Central and brachial BP will be concomitantly measured, with treating physicians, patients and investigators blinded towards allocation. As this trial is of a pragmatic design, all other aspects of BP and CKD management, including anti-hypertensive treatment-related decisions, diastolic BP targets, and clinical and laboratory follow-ups will be at the discretion of the attending Nephrologist. The primary outcomes include feasibility of large-scale trial using prespecified criteria and aortic stiffness (carotid-femoral pulse wave velocity) at 12 months. Other cardiovascular, renal, quality of life and safety outcomes will be evaluated.

Importance: CENTRAL-CKD is designed as a pilot trial aimed at providing the framework and justification to proceed to a large-scale trial with adequate power to detect the impact of the proposed intervention on clinically important outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age;
2. eGFR <30 mL/min/1.73m2 as determined by the CKD-EPI equation (within 30 days of screening);
3. Office brachial cuff systolic blood pressure between 120 and 160 mmHg (using automated office blood pressure).

Exclusion Criteria:

1. Already taking 5 or more anti-hypertensive medications (any class)
2. Unwillingness to change anti-hypertensive medication by the attending Nephrologist or patient
3. Recent acute kidney injury (>50% increase in serum creatinine in preceding 30 days)
4. Previous kidney replacement therapy (kidney transplant, hemodialysis or peritoneal dialysis)
5. Recent myocardial infarction, stroke, heart failure (in preceding 30 days)
6. Recent injurious fall requiring hospitalisation (in preceding 30 days)
7. Concomitant major illness / comorbidity that may result in death in the next 6 months
8. Participation in another study that is likely to affect BP levels
9. Inability to provide consent due to cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Consent rate | Baseline
  Proportion of participants who provide consent relative to the number approached for participation.
  Feasibility criteria (No / Probable / Yes): <30% / 30-60% / >60%
Feasibility: Recruitment rate | Baseline
  Proportion of randomized participants relative to the number of screened participants.
  Feasibility criteria (No / Probable / Yes): <40% / 40-80% / >80%
Feasibility: Achieved BP target rate | 12 months
  Proportion of randomized participants who achieve BP target at 12 months Feasibility criteria (No / Probable / Yes): <30% / 30-60% / >60%
Feasibility: Completion rate | 12 months
  Proportion of randomized participants who complete the trial Feasibility criteria (No / Probable / Yes): <40% / 40-80% / >80%
Feasibility: Recruitment pace | 12 months after activation of last site
  Number of participants recruited after 24 months of activation for all sites Feasibility criteria (No / Probable / Yes): <54 / 54-81 / >81
Feasibility: Divergent treatment decision rate | 12 months
  Proportion of divergent treatment decision based on central BP compared to brachial BP Feasibility criteria (No / Probable / Yes): <10% / 10-30% / >30%
Feasibility: Therapeutic inertia rate | 12 months
  Proportion of therapeutic inertia Feasibility criteria (No / Probable / Yes): >60% / 60-30% / <30%
Difference in aortic stiffness | 12 months
  Carotid-femoral pulse wave velocity

SECONDARY OUTCOMES:
Difference in eGFR decline | 12 months
Change in albuminuria | 12 months
Difference in Daily Defined Doses of blood pressure drugs | 12 months
Quality of life (KDQOL-SF questionnaire) | 12 months
  Score 0 to 100. Higher score represents better quality of life

OTHER OUTCOMES:
Progression towards kidney failure (sustained eGFR loss ≥ 40%, kidney replacement therapy initiation or death from renal failure) | 12 months
Major adverse cardiovascular adverse events (cardiovascular mortality, myocardial infarction, stroke, heart failure requiring hospitalisation, peripheral artery disease requiring revascularisation or amputation) | 12 months
  Composite and individuals outcomes
All-cause hospitalisation | 12 months
All-cause mortality | 12 months
Acute kidney injury (>50% increase in serum creatinine) | 12 months
Symptomatic orthostatic hypotension, dizziness, light headedness, injurious falls, syncope or any unexpected event attributable to the intervention | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Remi Goupil, MD MSc, Principal Investigator — Hôpital Sacré-Coeur de Montréal
Locations (1):
- Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goupil R, Nadeau-Fredette AC, Prasad B, Hundemer GL, Suri RS, Beaubien-Souligny W, Agharazii M. CENtral blood pressure Targeting: a pragmatic RAndomized triaL in advanced Chronic Kidney Disease (CENTRAL-CKD): A Clinical Research Protocol. Can J Kidney Health Dis. 2023 May 6;10:20543581231172407. doi: 10.1177/20543581231172407. eCollection 2023. PMID 37168686